CLINICAL TRIAL: NCT01110434
Title: Biobehavioral Effects of Topiramate on Cannabis-Related Outcomes in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Miranda, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01DA026778 (NIH); R01DA026778 (NIH)
Record Dates: First submitted 2010-04-20; First posted 2010-04-26 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Cannabis Abuse; Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): Topiramate (200 mg daily)
  Interventions: Drug: Topiramate
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate (200 mg daily)
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — Placebo (daily)
  Arms: Sugar pill

SUMMARY:
Cannabis use is a significant public health concern that disproportionately affect youth. Although promising psychosocial interventions are being developed, most youth do not benefit from these interventions alone. Given the clinical demand for effective treatments, the National Institute on Drug Abuse (NIDA) identified the critical need for data on the tolerability and potential efficacy of medications in adolescents. The purpose of this two-year study is to test if and how topiramate, a medication under intense study for treating several drugs of abuse, reduces cannabis use among teenagers. To this end, the investigators will randomize 56 nontreatment-seeking regular cannabis users (15 or 20 years old) to receive topiramate or placebo for 6 weeks. Youth will monitor their cannabis use for the 6-week period using handheld electronic diaries and complete assessments of reactivity to cannabis-related cues.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 20 years old (inclusive)
* Non-treatment seeking for cannabis abuse or dependence
* Able to read English, understand their rights as provided by the informed consent process, and be willing to sign an informed consent form to participant in the study
* If younger than 18 years old, informed consent from a parent or legal guardian is required
* Used cannabis at least 2 days per week during the past 30 days

Exclusion Criteria:

* Treatment seeking or a recent history of treatment for cannabis abuse or dependence
* Endorses a current commitment to stop using cannabis
* Clinically significant physical abnormalities as indicated by physical exam, hematological assessment, bilirubin concentration or urinalysis
* History of renal impairment, renal stones, seizures, or unstable hypertension
* Underweight (i.e., less than the 5th percentile) or overweight (equal to or greater than the 95th percentile), as determined by the Body Mass Index
* Positive urine toxicology screen for narcotics, amphetamines, or sedative hypnotics or self-reported drug use, other than cannabis, alcohol or nicotine, in the past 30 days
* Pregnant, nursing, or refusal to use reliable barrier method of birth control (e.g., condom), if female
* Took a psychotropic medication in the past 30 days
* Taking medications with a potential effect on cannabis use or a carbonic anhydrase inhibitor
* Suicidal
* A current DSM-IV-TR Axis I diagnosis other than attention- deficit/hyperactivity disorder or a disruptive behavior disorder
* A current substance use disorder other than a cannabis, alcohol, and nicotine use disorders
* Significant alcohol withdrawal symptoms
* Known sensitivity to topiramate

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miranda, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Meisel SN, Carpenter RW, Treloar Padovano H, Miranda R. Day-level shifts in social contexts during youth cannabis use treatment. J Consult Clin Psychol. 2021 Apr;89(4):251-263. doi: 10.1037/ccp0000647. PMID 34014688
- [Derived] Treloar Padovano H, Miranda R. Subjective cannabis effects as part of a developing disorder in adolescents and emerging adults. J Abnorm Psychol. 2018 Apr;127(3):282-293. doi: 10.1037/abn0000342. PMID 29672090

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Sugar Pill
Started | 40 | 26
Completed | 29 | 20
Not Completed | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Sugar Pill | Total
Number analyzed (Participants) | 40 | 26 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.30 (2.03) | 18.81 (2.08) | 19.71 (2.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 20 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Cannabis Use
Description: Frequency of Cannabis Use (Percent Use Days Per Week)
Time Frame: Weeks 1-6
Measure: Mean (Standard Deviation); unit: Percentage of use days
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 40 | 26
Percentage of use days | 55.89 (32.35) | 63.10 (34.91)

2. Secondary Outcome: Quantity of Cannabis Use
Description: Total Grams of Cannabis Use Per week
Time Frame: Weeks 1-6
Measure: Mean (Standard Deviation); unit: Grams Per Week
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 40 | 26
Grams Per Week | 1.87 (2.11) | 2.85 (3.29)

3. Secondary Outcome: Amount of Cannabis Use Per Use Day
Description: Average Grams of Cannabis Used Per Use Day
Time Frame: Weeks 1-6
Measure: Mean (Standard Deviation); unit: Average Grams Per Use Day
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 40 | 26
Average Grams Per Use Day | 0.46 (0.32) | 0.60 (0.48)

ADVERSE EVENTS:
Time Frame: Data were collected during the 6-week medication (or placebo pill) period.
Description: We followed the same definition as clinicaltrials.gov.
Arm/Group | Topiramate | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/26
Other Adverse Events (participants affected / at risk) | 35/40 | 24/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=40) | Sugar Pill (N=26)
Headache (General disorders) | 8 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Cough, Cold Symptoms (General disorders) | 5 | 5
Injury (General disorders) | 8 | 5
Parasthesias (General disorders) | 15 | 2
Sore Throat (General disorders) | 4 | 2
Runny Nose, Sinus Problems, Sneezing (General disorders) | 14 | 12
Stomach Pain, Cramps (Gastrointestinal disorders) | 2 | 3
Changes in Vision (Eye disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 12 | 8
Decrease in Appetite (General disorders) | 19 | 9
Weight Loss (General disorders) | 20 | 6
Irritability (Psychiatric disorders) | 2 | 3
Nervousness (Psychiatric disorders) | 4 | 0
Confusion (Psychiatric disorders) | 5 | 0
Difficulty with Coordination or Balance (General disorders) | 6 | 0
Difficulty with Memory (General disorders) | 8 | 5
Fatigue (General disorders) | 9 | 9
Anxiety (Psychiatric disorders) | 10 | 0
Depression (Psychiatric disorders) | 10 | 1
Dizziness (General disorders) | 10 | 2
Difficulty with Concentration or Attention (General disorders) | 11 | 2
Word Finding Difficulties (General disorders) | 11 | 4
Slow Thinking or Reactions (General disorders) | 12 | 4
Drowsiness or Sleepiness (General disorders) | 12 | 13
Fever (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No